CLINICAL TRIAL: NCT06570980
Title: Comparative Analysis of Cost-effectiveness Between Sulfonylureas and DPP4 Inhibitors in Combination With Metformin in Treatment of Type 2 Diabetic Patients : A Retrospective, Observational Study.
Status: Recruiting | Type: Observational
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Sheuly Akter, MD resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Other Study IDs: 4575
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM), Cost-effectiveness, Sulfonylureas, DPP4 Inhibitors, Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A- type 2 diabetic patients having sulfonylurease with metformin: Sulfonylurease- gliclazide(30/60/80mg), glimepiride (1/2/3/4mg), glibenclamide (5mg), glipizide (5mg)
  metformin - 500/850/1000mg
  Interventions: Drug: sulfonylurease with metformin, DPP4 inhibitors with Metformin
- Group B- type 2 diabetic patients having DPP4 inhibitors with metformin: DPP4 inhibitors- Linagliptin (2.5/5mg), Sitagliptin (50mg), Vildagliptin (50mg)
  metformin - 500/850/1000mg
  Interventions: Drug: sulfonylurease with metformin, DPP4 inhibitors with Metformin

INTERVENTIONS:
Drug: sulfonylurease with metformin, DPP4 inhibitors with Metformin — Oral hypoglycemic agents

SUMMARY:
The aim of this study is to compare the cost effectiveness of Sulfonylureas and DPP4-inhibitors in combination with Metformin among type2 diabetic patients diagnosed for 2-5 years. Glycemic status and other clinical outcome are compared in between two groups and ICER are compared.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a highly prevalent chronic disease. Every 3 in 4 adults have diabetes in low and middle income countries. Diabetes costs about 966 billion USD dollars in total health expenditure. This is a huge economic burden for low and middle income countries, where people have to pay out of their pocket for medical expense. Type2 Diabetes is responsible for various serious life threatening complications like cardiovascular death, retinopathy, nephropathy, stroke etc.

Along with diet and exercise, lifelong pharmacotherapy is needed. But cost of drug is increasing day by day, especially newer agents are very much expensive. The aim of this study is to compare the cost and effectiveness of Metformin plus sulfonylureas with Metformin plus DPP4 inhibitors in management of type 2 diabetic patient. This research will be conducted in Pharmacology department of Bangabandhu Sheikh Mujib Medical University (BSMMU), outpatient department of BIRDEM General Hospital, and Siddhirganj diabetic center, Narayanganj from the day of approval by IRB to July, 2024. It will be multi centered, retrospective, observational, cost-effectiveness study. It will involve type 2 diabetic patients who have diagnosed for 2 years and taking either any of sulfonylurease or DPP4 inhibitors along with Metformin. 206 patients will be enrolled, 103 in each group. One group will who are taking sulfonylureas with Metformin and another group will who are taking DPP4 inhibitors with Metformin. Primary outcome will be glycemic control which will be measured by HbA1c % and secondary outcome will be cardiovascular events like hypertension, angina, myocardial ischemia for which ECG and patients medical record will be analyzed, nephropathy will be classified by eGFR, insulin therapy and any hospitalization needed or not. Data will be collected about various socio-demographic variables such as age, sex, education, family history of diabetes, other co morbidities. Hypertension with diabetes will be considered in equal percentage in both groups. Total direct medical cost like drug price, hospitalization and cost of adverse drug reaction will be measured which will be actual medical cost of individual patient. Then cost-effectiveness analysis will be done by ICER. Descriptive statistics will be used for demographic variables. Means & standard deviation for ii continuous variables and number & percentage for categorical variables will be used. T test can be used to compare cost in two groups. Chi-square test may be used to compare clinical outcome. Price of drug will be obtained from BDNF 5th edition for particular brand of above mentioned drug in every individual patient. This study will revealed whether there is significant difference in healthcare costs and clinical outcome between the above mentioned two groups. This retrospective study will provide valuable insight about cost effectiveness of sulfonylureas and DPP4 inhibitors for the management of T2DM. Healthcare providers even policymakers can be benefitted to take informed decision in patient care and formulary choices.

ELIGIBILITY:
Inclusion Criteria:

* New onset type2 diabetes mellitus diagnosed for 2 -5 years.
* Taking either sulfonylurea or DPP4 inhibitors combined with Metformin from the time of diagnosis.
* Age 18 years or above.
* Both male and female.
* Provided written informed consent.

Exclusion Criteria:

* Unwillingness to participate or unwillingness to give written informed consent.
* Patients on Insulin therapy or monotherapy with metformin since the time of diagnosis.
* Taking other than sulfonylurea or DPP4 inhibitors combined with Metformin from the time of diagnosis.
* Diabetes related complications at the time of diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending out patient department of BIRDEM General hospital,Shahbag, Dhaka, which is a tertiary care hospital and patients attending Siddhirganj Diabetic center, a secondary care level diabetes center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c% | 2-5years
  achievment of target HbA1 less than 7%

SECONDARY OUTCOMES:
Insulin therapy | 2-5years
  requirement of insulin therapy
hospitalization | 2-5years
  requirement of hospitalization
3rd line therapy | 2-5years
  addition of any 3rd drug
nephropathy | 2-5years
  development of nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sheuly Akter, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes